CLINICAL TRIAL: NCT01461408
Title: Promoting HPV Vaccination Through African American Beauty Salons: a Pilot Test of a Culturally-Competent Education and Empowerment Strategy
Brief Title: Promoting Human Papillomavirus (HPV) Vaccination Through African American Beauty Salons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MEE Productions, Inc. (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Ivan Juzang, President, MEE Productions, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Merck-IISP-39187
Record Dates: First submitted 2011-10-13; First posted 2011-10-28 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Human Papilloma Virus
Keywords: HPV Vaccination; Beauty Salons; Health Education; Sexual Health
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (16):
- Beauty Salon #1b (Experimental): Females ages 18-26
  Interventions: Behavioral: Health Education Session
- Beauty Salon #1a (Experimental): Mothers of 9-18 year old females
  Interventions: Behavioral: Health Education Session
- Beauty Salon #2b (Experimental): Females ages 18-26
  Interventions: Behavioral: Health Education Session
- Beauty Salon #3a (Experimental): Mothers of 9-18 year old females
  Interventions: Behavioral: Health Education Session
- Beauty Salon #3b (Experimental): Females ages 18-26
  Interventions: Behavioral: Health Education Session
- Beauty Salon #4a (Experimental): Mothers of 9-18 year old females
  Interventions: Behavioral: Health Education Session
- Beauty Salon #4b (Experimental): Females ages 18-26
  Interventions: Behavioral: Health Education Session
- Beauty Salon #2a (Experimental): Mothers of 9-18 year old females
  Interventions: Behavioral: Health Education Session
- Beauty Salon #5a (Experimental): Mothers of 9-18 year old females
  Interventions: Behavioral: Health Education Session
- Beauty Salon #5b (Experimental): Females ages 9-26
  Interventions: Behavioral: Health Education Session
- Beauty Salon #6a (Experimental): Mothers of 9-18 year old females
  Interventions: Behavioral: Health Education Session
- Beauty Salon #6b (Experimental): Females ages 18-26
  Interventions: Behavioral: Health Education Session
- Beauty Salon #7a (Experimental): Mothers of 9-18 year old females
  Interventions: Behavioral: Health Education Session
- Beauty Salon #7b (Experimental): Females ages 18-26
  Interventions: Behavioral: Health Education Session
- Beauty Salon #8a (Experimental): Mothers of 9-18 year old females
  Interventions: Behavioral: Health Education Session
- Beauty Salon #8b (Experimental): Females ages 9-18
  Interventions: Behavioral: Health Education Session

INTERVENTIONS:
Behavioral: Health Education Session — The educational messages during the education session will engage individual women, their peer group, their family members and community influencers in a way that is authentic and share-able. Involving women in give-and-take discussions with people they trust and respect-their hairdressers-will be essential to increasing the number of them who consider the HPV vaccine for themselves and for those they care about.
  The investigators plan to recruit eight (8) predominantly African American beauty salons in Philadelphia and train multiple stylists in each salon to act as in-salon educators and facilitators for client recruitment to sexual health education sessions. These education sessions will be run by trained health educators (also African American females) and take place during "down times" in each of the salons, on a rotating basis. There will be two types of sessions offered, one for mothers of females ages 9-18 and one for females ages 18-26.

SUMMARY:
The investigators propose a non-randomized pilot study to assess the feasibility and effectiveness of using urban beauty salons as settings for culturally-competent health education about HPV vaccination. The educational messages will engage individual women, their peer group, their family members and community influencers in a way that is authentic and share-able. Involving women in give-and-take discussions with people they trust and respect-their hairdressers-will be essential to increasing the number of them who consider the HPV vaccine for themselves and for those they care about. The investigators believe that it is only after women who are opinion leaders among their peers begin positively supporting HPV prevention that it will gain wider acceptance.

The investigators plan to recruit eight (8) predominantly African American beauty salons in Philadelphia and train multiple stylists in each salon to act as in-salon educators and facilitators for client recruitment to sexual health education sessions. These education sessions will be run by trained health educators (also African American females) and take place during "down times" in each of the salons, on a rotating basis.

* The investigators hypothesize the ability to successfully recruit eight (8) beauty salons for participation
* The investigators hypothesize the ability to successfully train multiple stylists per site to talk to their clients about HPV and its impact on women of color
* The investigators hypothesize that knowledge and awareness of HPV, as well as intentions to vaccinate will significantly improve among women who attend a salon-based health education session

ELIGIBILITY:
Inclusion Criteria:

* Mother of an 9-18 year old female
* Female who is 18-26 years old

Exclusion Criteria:

* Not a mother of an 9-18 year old female
* Not a female who is 18-26 years old

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Recruitment of 8 beauty salons | 6 months
  To recruit 8 beauty salons from Philadelphia PA that would be willing to have their stylists trained to be part of the study, as well as have their salon serve as a host site for education sessions for their female customers.

SECONDARY OUTCOMES:
Intentions to Vaccinate Against HPV | 18 months
  To increase knowledge and awareness about HPV, as well as intentions to vaccinate among beauty salon clients. Intentions to vaccinate will be measured with a single item using the following wording "How likely are you (or your daughter) to start the HPV vaccine series in the next 6 months?". Response options range from "very likely" to "very unlikely" using a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Juzang, MBA, Principal Investigator — MEE Productions, Inc.; Amy Leader, DrPH, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Pre-selected beauty salons, Philadelphia, Pennsylvania, United States